CLINICAL TRIAL: NCT03665779
Title: Nitric Oxide Donor Isosorbide Mono Nitrate for Cervical Ripening in Induction of Labor in Term or Post Term Pregnancies in Females With Pre-labor Rupture of Membranes
Brief Title: Nitric Oxide Donor Isosorbide Mono Nitrate for Induction of Labor With Pre-labor Rupture of Membranes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ahmed nagy shaker ramadan (Other)
Responsible Party: Sponsor-Investigator, ahmed nagy shaker ramadan, resident of obstetrics and gynecology, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AN1988
Record Dates: First submitted 2018-08-30; First posted 2018-09-11 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Induction of Labor Affected Fetus / Newborn; Rupture of Membranes Prior to Onset of Labor
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — isosorbide-5-mononitrate; Pyridoxine

STUDY DESIGN:
Intervention Model Description: The patients will be divided into 2 groups:
  Group 1:
  70 pregnant females, induction of labor will be done by Intra vaginal isosorbide mono nitrate (Effox 40 mg MINAPHARM)
  Group 2:
  70 pregnant females, induction will be done by placebo (pyridoxine) administered in the posterior vaginal fornix.
Who Masked: Participant, Investigator
Masking Description: A double-blind study is one in which neither the participants nor the experimenters know who is receiving a particular treatment. This procedure is utilized to prevent bias in research results. Double-blind studies are particularly useful for preventing bias due to demand characteristics or the placebo effect. In a double-blind study, the investigators who interact with the participants would not know who was receiving the actual drug and who was receiving a placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isosorbide mono-nitrate group (Experimental): 70 pregnant females, induction of labor will be done by Intra vaginal isosorbide mono nitrate (Effox 40 mg MINAPHARM)
  Interventions: Drug: isosorbide mononitrate
- placebo group (Placebo Comparator): 70 pregnant females, induction will be done by placebo (pyridoxine) administered in the posterior vaginal fornix.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: isosorbide mononitrate — 70 pregnant females, induction of labor will be done by Intra vaginal isosorbide mono nitrate (Effox 40 mg MINAPHARM) repeated every 4 hours maximum 4 times
  Other Names: Effox
  Arms: isosorbide mono-nitrate group
Drug: Placebo — 70 pregnant females, induction will be done by placebo (pyridoxine) administered in the posterior vaginal fornix.repeated every 4 hours maximum 4 times
  Other Names: pyridoxine
  Arms: placebo group

SUMMARY:
The study aims to evaluate and assess the effectiveness and safety of vaginal administration of isosorbide mono nitrate (IMN) to induce cervical ripening and shorten the interval time between induction and delivery in women undergoing induction of labor at term or post term with prelabor rupture of membrane.

Research Hypothesis:

In women undergoing induction of labor at term or post term with pre-labor rupture of membrane, vaginal administration of isosorbide mono nitrate (IMN) is effective to induce cervical ripening and shorten the interval time between induction and delivery.

Research Questions:

Does vaginal administration of isosorbide mono nitrate (IMN) induce cervical ripening and shorten the interval time between induction and delivery in women undergoing induction of labor at term or post term with prelabor rupture of membrane?

DETAILED DESCRIPTION:
* Study Design: Prospective double blinded randomized placebo-controlled Clinical trial
* Time plan: Approximately 6 months according to calculated sample size.
* study setting: this study will be conducted obstetrics and gynecology department at Cairo university.
* study population: patient will be recruited in this study those attending labor ward for induction of labor in term or post term pregnancies in females with pre-labor rupture of membranes
* Methodology in details

All women will be subjected to

-History taking:

* Verbal consent.
* Detailed clinical history.
* Personal history: Name, Age, Parity, Occupation, Residency and Special habits.
* Present history: History of onset, course and duration of vaginal bleeding or bloody vaginal discharge, presence of uterine contraction, PROM, IUGR or any indication of induction of labor.
* Obstetric history: History of previous preterm labor, previous abortion, previous full term deliveries, RH incompatibility, mode of delivery and fetal outcome.
* Menstrual history: For estimation of gestational age using Naegele's rule, provided that she had regular cycles for the last three months before she got pregnant and was not taking contraceptive pills during this period and she was sure of her dates.

Term pregnancy defined as delivery between 37 and 42 weeks of gestation. Gestational age was assessed from the menstrual history and confirmed by measurement of fetal crown-rump length at a first-trimester scan. Post-term pregnancy defined as delivery after 42 weeks of gestation.

* Past history: History of medical disorders, drug therapy or allergy or history of intake of other tocolytic drugs.
* Family history : For any similar condition

  -Examination
* Full clinical examination (pulse, temperature and the blood pressure).
* General examination including chest, heart and abdominal examination for fundal level.
* Local clinical examination; with special attention to pelvic examination to assess the state of the cervix (dilatation, effacement, PROM, station and presenting part) and to assess vaginal bleeding or amniotic fluid in vagina if present and to exclude cephalic-pelvic disproportion.
* Routine ante-natal investigations (Rh, Hb, fasting and postprandial blood sugar and complete urine analysis).(CBC with differential and CRP to exclude chorioamnionitis)
* Ultrasonography examination : to assess the following data:
* Gestational age
* Fetal viability
* Fetal presentation and EFW.
* Exclusion of any fetal congenital anomalies.
* To ensure that the all inclusion criteria are present.
* Check amniotic fluid index.

  * Intervention:

After admission for labor induction, cervical assessment is done to see dilatation (cm), length (cm), position, consistency, and station of presenting part to get the modified Bishop score and to confirm pre-labor rupture of membrane.

In vaginal IMN group (group 1) 40 mg tablet of intra-vaginal IMN (Effox; MINAPHARMA, Cairo, Egypt) will be placed into the posterior fornix of the vagina, through a digital vaginal examination, every 4 h for a maximum of four doses. The medication will be stopped with the onset of labor. Oxytocin will be started 6 h after the last dose of IMN in women not in active phase of labor but have Bishop score is >6. Intravenous oxytocin is initiated at an infusion flow rate of 4 mIU/min and will be doubled as necessary, with 30-min intervals between increasing the doses, up to a maximum of 16 mIU/min. To obtain this concentration, 5 IU of synthetic oxytocin are added to 500 ml of a 5% dextrose solution. Further management of labor will be done according to the hospitals protocols.

In placebo group (group 2) 40 mg intra-vaginal pyridoxine placebos every 4 h for a maximum of four doses will be given, followed by intravenous oxytocin infusion and management of labor as in group 1.

In both groups, the pregnant females who don't progress to labor (regular contractions with continued cervical changes) with no cervical changes ( bishop score equal to or less than 6) after a maximum of four doses and oxytocin infusion, this will be considered failure of induction and those patients will delivered by cesarean section.

Subjects will be followed-up regularly after taking the medications by obstetricians who are unaware of the group to which the patient belongs. Uterine contraction and fetal heart rate (FHR) will be checked every 30 min. Prophylactic or "latency" antibiotics, typically ampicillin and erythromycin for prevention of chorioamnionitis. Symptoms and vital signs will be monitored at regular intervals. Subjects will be asked to report when they have uterine contraction or abnormal symptoms such as headache, nausea, shivering.

signs of chorioamnionitis (e.g : fever, uterine fundal tenderness, maternal and fetal tachycardia, purulent or foul smelling discharge) will be checked at regular intervals.

Pelvic examination will be done with each dose and with the onset of uterine contractions. Doses will be stopped with the onset of uterine contractions or when the maximum doses reached.

After documentation of all the collected data, the following will be studied:

* Induction to onset of labor time.
* Induction to delivery time.
* Failure of induction due to maternal or fetal cause.
* Need for augmentation of labor by oxytocin.
* Recording any maternal or fetal morbidities.

Possible Risk:

Risks of induction of labor as failure of induction or maternal or fetal morbidities.

Side effects of the used drugs. Complications of PROM either maternal or fetal.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.
* Cephalic presentation.
* Bishop score < or = 6.
* Average size of the fetus.
* Adequate pelvic dimensions.
* Prelabour rupture of membranes.
* Term or post-term pregnancies with an indication for labor induction either maternal or fetal.

Exclusion Criteria:

* Previous uterine scar (e.g. caesarian delivery or unknown uterine incision , previous hysterotomy or myomectomy of the uterine corpus involving entry of the uterine cavity or extensive myometrial dissection, previous uterine rupture)
* Patients with regular uterine contractions.
* Malpresentation.
* Multifetal gesta1tion.
* Established fetal distress ( e.g. thick meconium stained liguor or non reassuring CTG changes)
* Indication for CS, e.g. Major degree of cephalopelvic disproportion and fetal macrosomia.
* Placenta previa or vasa previa.
* Active genital herpes infection.
* Severe maternal illness (e.g. severe preeclampsia).
* Laboratory and clinical sign of chorioamnionitis.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 140 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
induction of labor | up to 24 hours
  the effectiveness and safety of vaginal administration of isosorbide mono nitrate (IMN) to induce cervical ripening for induction of labor at term or post term pregnancy with prelabor rupture of membrane regarding (Induction to onset of labor time, Induction to delivery time)

CONTACTS AND LOCATIONS:
Overall Officials: waleed M EL Khyat, MD, Principal Investigator — university
Locations (1):
- faculty of medicine - Cairo university, Cairo, Kasr El Ainy, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Afifi AN, Taymour MA, El-Khayat WM. Isosorbide mononitrate for cervical ripening in induction of labor for pregnant women with PROM at or post term. Int J Gynaecol Obstet. 2021 Dec;155(3):512-517. doi: 10.1002/ijgo.13604. Epub 2021 Feb 18. PMID 33458819